CLINICAL TRIAL: NCT02855021
Title: Prediction of Dementia in Parkinson's Disease by Measuring Cerebral Metabolism With PET Scan
Acronym: PREDEMPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P140306
Record Dates: First submitted 2016-06-27; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Parkinson Disease
Keywords: Dementia; Cerebral metabolism; PET scan
MeSH Terms: conditions — Parkinson Disease; Dementia | interventions — Space Flight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parkinson disease (Other): Patients with a Parkinson disease with clinical diagnosis made for at least 5 years
  Interventions: Other: Explorations

INTERVENTIONS:
Other: Explorations — Imaging tests and neuropsychological assessment are carried out within 60 days following patient enrollment.
  Neuropsychological assessment lasts 1:30 to 2:00 hours and is conducted by a psychologist in an interview during which patient will pass several tests on memory, language, attention or orientation in space.
  These tests do not require discontinuation of Parkinson's disease treatment.

SUMMARY:
Parkinson's disease (PD) is a common disease. Dementia will affect 80% of these patients during their evolution. In addition, treatments of motor signs have a potential impact on these disorders and conversely.

The purpose of this study is to show focal abnormalities in brain metabolism in the precuneus and posterior cingulate region are predictive of the onset of dementia within 2 years.

DETAILED DESCRIPTION:
Cognitive impairment and dementia have become major factors of disability induced by Parkinson's disease. The prediction of dementia in any given patient may be useful for prognosis but also for discussion of setting up heavy therapeutic techniques, especially surgical. Currently, known predictors are disease severity, age and existence of pre-cognitive disorders; other assumptions are discussed. Among these, morphological imaging techniques (MRI) and functional techniques (MRI, PET) are proposed.

Use increasingly early of heavy, expensive and potentially ineffective surgical treatment in dementia makes it necessary to find independent, early and reliable markers of the onset of dementia in Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria

* Male or female with Parkinson's Disease
* 45 < Age ≥ 75 years
* Parkinson's disease with clinical diagnosis made for at least 5 years (60 months)
* Patient able to perform cognitive tests in French during 1 hour 30 minutes
* Patient having provided a signed consent to participate in this trial
* Be either affiliated to, or a beneficiary of, a social security category
* Existence of caregiver at least contactable by phone

Exclusion Criteria

* Parkinson's disease diagnosed before 40 years old
* Clinical evidence for dementia or dementia criteria according to level 1 MDS-Task Force (Dubois et al. 2007)
* Atypical form of parkinsonism
* Other disease affecting the central nervous system
* Poorly controlled diabetes with glucose > 2.0 g/l or HbA1c>7,5% based on results of less than 3 months
* Taking a cholinesterase inhibitor treatment, memantine or long-term benzodiazepines other than referred hypnotic, neuroleptic
* History of surgery for Parkinson's disease or planned surgery within 6 months. Surgery is possible beyond
* Cons-indication to 3T MRI
* Inability to lie down for 60 minutes
* Legal protection
* Patient living outside the Ile-de France region

Secondary exclusion criteria

* Pregnant, breastfeeding or non-menopausal woman not taking contraception in the first 2 months of the study
* Existence of a significant brain injury on MRI
* Neuropsychological assessment at baseline showing dementia
* Fasting glucose > 1.6 g/l the day of FDG-PET

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Onset of dementia authenticated by a neuropsychological assessment (MDS Task Force criteria) | Year 2

SECONDARY OUTCOMES:
Regional cerebral glucose consumption in the parietal lobes studied with fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) and regional glucose consumption in the caudate nucleus and prefrontal areas studied with FDG PET | Day 90
Determination of cerebral blood flow (CBF) by arterial spin labelling (ASL) perfusion 3Tesla (3T) Magnetic Resonance Imaging (MRI) | Day 90
Identifying different striatal functional connectivity patterns by resting state functional MRI at 3T | Day 90
Cerebral cortex trophicity by VBM technique (Voxel-based morphometry) | Day 90
Number of hyperintensities in the FLAIR MR image | Day 90
Concentration of iron in the mesencephalon measured with MRI | Day 90
Degree of anosmia measured with the University of Pennsylvania Smell Identification Test (UPSIT) | Day 90
Correlation between initial clinical, neuropsychological and biological parameters and risk of onset of dementia | Day 0 and year 2

CONTACTS AND LOCATIONS:
Overall Officials: Claire THIRIEZ, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided